CLINICAL TRIAL: NCT07324174
Title: A Randomized Controlled Trial on the Effectiveness of Early Versus Conservative Rehabilitation Following Rotator Cuff Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Collins Ogbeivor, Clinical Consultant Physical Rehabilitation, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#2251676
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear, post rotator cuff repair, physical rehabilitation, early rehabilitation, delayed rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Exercise Therapy; Educational Status; Counseling; Control Groups

STUDY DESIGN:
Intervention Model Description: From the day after surgery, participants in the intervention group will engage in supervised passive range of motion (ROM) exercises focusing on forward flexion and external rotation. They will receive daily instructions for table slides and active movements for the elbow, wrist, and hand, while practicing passive shoulder flexion and abduction within their pain limits. Gentle pendulum exercises and passive movements are encouraged three times daily to improve shoulder mobility. Active shoulder exercises will be restricted until six weeks post-surgery to ensure proper healing. Sling use will gradually decrease by the sixth week, allowing active ROM exercises to begin. The control group will follow a delayed rehabilitation protocol with strict sling immobilization for the first six weeks, only allowing sling removal for basic exercises and activities. After six weeks, they will also start active ROM exercises.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Participants in the control group will follow a delayed rehabilitation protocol, learning strict sling immobilization techniques for the first six weeks postoperatively. During this period, sling removal will be allowed only for basic exercises and daily activities, with no other shoulder movements encouraged initially. Sling use will end by the sixth week, followed by the start of active ROM exercises.
  Interventions: Other: Group B (Control Group)
- Intervention arm (Experimental): From the day after surgery, the intervention will engage in supervised passive range of motion (ROM) exercises, focusing on forward flexion and external rotation. They will receive daily exercise instructions, including table slides and active movements for the elbow, wrist, and hand, while also practicing passive shoulder flexion and abduction based on their pain limits. Participants are encouraged to do gentle pendulum exercises and passive movements three times daily to improve shoulder mobility. Active shoulder exercises will be restricted until six weeks post-surgery to ensure healing. Sling use will decrease by the sixth week, allowing for active ROM exercises to start.
  Interventions: Other: Group A; Other: Therapeutic exercises, education and advice

INTERVENTIONS:
Other: Group A — From postoperative Day 1, participants will perform passive range of motion (ROM) exercises twice daily under the guidance of a physical therapist, focusing on forward flexion and external rotation. They will also receive instructions to perform specific daily exercises, including table slides, active elbow, wrist, and hand movements, and passive shoulder flexion and abduction-all within the limits of pain. Outside of these structured sessions, gentle pendulum exercises and additional passive movements (including abduction, flexion, and external rotation to 30 degrees) will be recommended three times daily to promote ROM and shoulder mobility. Active shoulder exercises will be restricted until postoperative week 6. Sling use will be gradually discontinued by week 6, at which point active-assisted ROM will be introduced. Full active ROM will be targeted by week 12, followed by progression to strengthening exercise.
  Other Names: Therapeutic exercises; Education and advice
  Arms: Intervention arm
Other: Therapeutic exercises, education and advice — Intervention will be provided with passive exercises and education from day one after surgery.
  Arms: Intervention arm
Other: Group B (Control Group) — Participants in the control group will follow a delayed rehabilitation protocol, learning strict sling immobilization techniques for the first six weeks postoperatively. During this period, sling removal will be allowed only for basic exercises and daily activities, with no other shoulder movements encouraged initially. Sling use will end by the sixth week, followed by the start of active ROM exercises.
  Other Names: Education and Advice
  Arms: Control arm

SUMMARY:
Background Rotator cuff tears (RCTs) are a common, costly, and often persistent musculoskeletal complaint, with an increasing number of shoulder pain patients undergoing surgical repair each year. Whereas many asymptomatic RCTs can be successfully managed non-surgically, when conservative treatment fails, surgery is recommended. However, there is a lack of consensus on the best approach to postoperative rehabilitation, an important factor in the recovery process of rotator cuff repairs. This study aims to investigate the effectiveness of early versus delayed rehabilitation following rotator cuff repairs.

Objective This study aims to determine the effectiveness of early versus delayed rehabilitation following rotator cuff repairs.

Method A two-armed, randomized controlled trial will be conducted in an outpatient physical rehabilitation department at a tertiary hospital. The sample will include 88 adults aged 18 years or older with RCTs. From the day after surgery, the intervention will engage in supervised passive range of motion (ROM) exercises, focusing on forward flexion and external rotation. They will receive daily exercise instructions, including table slides and active movements for the elbow, wrist, and hand, while also practicing passive shoulder flexion and abduction based on their pain limits. Participants are encouraged to do gentle pendulum exercises and passive movements three times daily to improve shoulder mobility. Active shoulder exercises will be restricted until six weeks post-surgery to ensure healing. Sling use will decrease by the sixth week, allowing for active ROM exercises to start. Participants in the control group will follow a delayed rehabilitation protocol, learning strict sling immobilization techniques for the first six weeks postoperatively. During this period, sling removal will be allowed only for basic exercises and daily activities, with no other shoulder movements encouraged initially. Sling use will end by the sixth week, followed by the start of active ROM exercises.

Outcome measures will include shoulder ROM, muscle power, a numeric pain scale (NPS), shoulder pain disability index (SPADI), and EQ-5D-5L questionnaires assessed at 3, 6, and 12 months follow-up between the two groups. Rotator cuff integrity will be evaluated using MRI at baseline and at 12 months post-surgery.

Conclusion We anticipate that this study will add to the body of knowledge required to make effective treatment choices on the management of patients following rotator cuff repairs. Ultimately, this trial aims not only to influence national rehabilitation guidelines but also to enrich the global evidence base concerning optimal rehabilitation strategies following rotator cuff repair, especially for populations in the Middle East and Gulf regions.

DETAILED DESCRIPTION:
Introduction Shoulder pain affects one in three people at some point in their lives (Chester et al., 2013; van der Heijden, 1999). It is one of the most common musculoskeletal conditions, with an estimated lifetime prevalence of up to 70% (Cadogan et al., 2011; Carr et al., 2015). The leading cause of shoulder pain and disability is rotator cuff tears (RCTs) (Largacha et al., 2006; Flatow et al., 1994). RCTs are a frequent and costly problem that often results in persistent pain, with more patients choosing surgical repair each year (Sealey and Lewis, 2016). Many asymptomatic RCTs can be effectively managed non-surgically through physiotherapy-led exercises, pain medications, or cortisone injections. However, when conservative treatments fail, surgical intervention may be recommended. While both surgical and non-operative treatments have their risks and benefits, a significant percentage of individuals have asymptomatic RCTs. Over time, many of these patients are at risk of developing symptoms of pain and disability (Tashjian, 2012).

Using high-resolution sonography, Yamaguchi et al. (2001) studied 58 patients with unilateral symptomatic full-thickness RCTs alongside a contralateral asymptomatic tear. They found that 51% of the previously asymptomatic tears developed pain symptoms and showed reduced shoulder function over a mean follow-up period of 2.8 years. Additionally, 50% of the newly symptomatic tears increased in size, while only 20% of the asymptomatic tears progressed. This study indicates that if RCTs are left unrepaired, they have limited capacity for self-healing. More importantly, it suggests a significant risk of tear progression, which correlates with increased shoulder pain and loss of function. Furthermore, Mall et al. (2010) conducted a prospective study involving a cohort of 195 patients diagnosed with asymptomatic RCT (RCTs). This study examined the progression of pain, shoulder function, and tear size over time. The researchers compared 44 patients who developed symptoms to a matched group of 45 who remained asymptomatic. The findings revealed that individuals with asymptomatic RCTs who became symptomatic experienced a substantial decline in shoulder function and an increase in tear size, showing a 23% increase compared to only 4% for those who remained asymptomatic, approximately two years after the initial evaluation (P < 0.1) Previous studies (Maman et al., 2009; Safran et al., 2011) have indicated that patients with symptomatic full-thickness tears who undergo conservative treatment face a significant risk of experiencing an additional 50% tear within two years. Consequently, early surgical intervention is advised for young adults (aged 65 and younger) with significant (> 1-1.5 cm) reparable full-thickness tears, provided they do not exhibit chronic muscle changes, due to the increased likelihood of developing a larger tear over time (Tashjian, 2012). Additionally, surgical repair is recommended for acute RCT across all age groups, except for those with small (< 1-1.5 cm) full-thickness tears. This recommendation is based on the substantial risks of irreversible changes associated with conservative treatment and the high probability of healing when repair is performed promptly (Mantone et al., 2000). For instance, Petersen and Murphy (2011) suggest that substantial (> 1-1.5 cm) acute full-thickness tears should ideally be repaired within three weeks of the injury to maximize the restoration of shoulder function.

Clinical studies (Weber, 1999; Kartus et al., 2006) evaluating patients with partial-thickness and full-thickness RCTs have shown that those treated with arthroscopic debridement and acromioplasty, without tendon repair, exhibited limited spontaneous healing of the rotator cuff. Prospective longitudinal studies indicate that the long-term clinical outcomes for both arthroscopic and open rotator cuff repairs are favorable, with over 90% of patients reporting good or excellent results at a 10-year follow-up (Galatz et al., 2001; Wolf et al., 2004). However, the effectiveness of these surgical interventions can vary depending on factors such as the patient's age, the extent of the tear, and the presence of any comorbid conditions.

Further research is needed to identify optimal treatment strategies that can enhance healing and improve functional outcomes for patients with RCTs following surgery. Additionally, exploring the role of rehabilitation protocols and postoperative care may provide valuable insights into maximizing recovery and minimizing the risk of re-tears. In practice, most post-surgical rehabilitation protocols for RCT repairs focus on protecting the repaired tissue, strengthening the rotator cuff and scapulothoracic muscles, and improving shoulder range of motion [ROM] (Corban et al., 2024). However, there remains a debate regarding the most effective rehabilitation protocol for post-surgery RCT patients.

Rehabilitation typically takes between 4 and 12 months, with patients often immobilized in a sling for 4 to 6 weeks after surgery (Sheps et al., 2018). Nevertheless, there is conflicting evidence regarding the optimal duration of postoperative immobilization (Chang et al., 2015; Chan et al., 2014). Some authors suggest that early mobilization may reduce patient burden and the occurrence of postoperative shoulder stiffness and muscle atrophy but may also increase the risk of re-tears (Chang et al., 2015; Papalia et al., 2012; Denard et al., 2011). Tirefort et al. (2019), in a well-designed randomized controlled trial, compared clinical and radiographic outcomes for up to 6 months post-rotator cuff repair with and without postoperative sling immobilization in a cohort of 80 patients with isolated full-thickness superior small to medium-sized RCTs. The study found that patients who did not use a sling had better outcomes, including reduced shoulder pain, improved mobility, and higher functional scores, compared to those who underwent sling immobilization at the 3 and 6-month follow-ups. However, due to the small sample size of the participants, the findings of this study should be interpreted cautiously. A systematic review conducted by Mazuquin and colleagues (2018) examined the effectiveness of early rehabilitation compared to conservative rehabilitation for patients who underwent postoperative repair of rotator cuff tears (RCTs). The study found no significant differences in shoulder function, pain levels, ROM (ROM), or rates of retears between the two approaches. Nonetheless, the authors concluded that early mobilization might be advantageous, especially for small and medium tears, and they called for additional high-quality research, including larger randomized controlled trials (RCTs).

More recently, in a systematic review and meta-analysis, Mazuquin et al. (2021) further explored the effectiveness of early versus delayed rehabilitation for patients who have received RCT repair. The study encompassed twenty randomized controlled trials involving a total of 1,841 patients. The authors noted significant variations in the rehabilitation protocols, including the timing of sling use and the progression of exercises. They highlighted that despite rotator cuff repair being a common surgical procedure, postoperative rehabilitation practices have largely remained unchanged for over two decades. The findings from their review indicated that patients who engaged in early rehabilitation may achieve a greater ROM sooner without increasing the risk of compromising the repair integrity-an ongoing concern for clinicians, especially shoulder orthopedic surgeons. The authors urged the need for a large, high-quality randomized controlled trial that encompasses all sizes of RCTs, emphasizing a more progressive and individualized approach to early rehabilitation. This approach should involve a gradual introduction of active arm use as soon as feasible, always within the limits of the individual patient's pain tolerance. This is the motivation of this current study. This study aims to evaluate the effectiveness of early versus delayed rehabilitation following rotator cuff repairs.

Objective and Hypotheses The primary objective of this randomized controlled trial (RCT) is to assess the effectiveness of early rehabilitation compared to delayed rehabilitation in patients who have undergone rotator cuff tear (RCT) repair. The hypothesis posits that early rehabilitation will result in superior outcomes concerning shoulder pain and function when compared to the conservative approach.

Research Question Is early rehabilitation more effective in enhancing shoulder outcomes post-RCT repair than delayed rehabilitation?

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older
2. Patients diagnosed with a symptomatic tear of the rotator cuff and listed for surgical repair
3. Rotator cuff tear confirmed by MRI
4. Patients screened by the surgeon as suitable to participate
5. Able to attend out-patient follow-up physiotherapy appointment
6. Demonstrate the ability and willingness to consent and continue participation in the study
7. Able to understand Arabic or English Language

Exclusion Criteria:

A patient will not be eligible for participation in the study if any of the following criteria apply:

1. Individuals younger than 18 years
2. Those unable or unwilling to consent or continue with the study.
3. Moderate to severe arthritis seen on x rays or MRI
4. Fatty infiltration grade >= 3

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male and female genders
Enrollment: 86 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability score | From enrollment to the end of study at 12 months
  The Shoulder Pain and Disability Index (SPADI) will be used to evaluate potential participants' shoulder pain and function. This self-report questionnaire assesses pain and disability related to musculoskeletal shoulder issues [39]. SPADI consists of 13 items divided into two domains: pain (5 questions) and disability (8 questions), scored from zero (no pain or difficulty) to ten (worst pain or difficulties needing assistance). Each domain equally contributes to an overall percentage score, with zero indicating no issues and 100% indicating maximum pain and disability. It will be measured by a trained, experienced and quality physical therapist at baseline, 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
This is not supported by the hospital IRB requirements.

REFERENCES:
- [Background] Mazuquin B, Moffatt M, Gill P, Selfe J, Rees J, Drew S, Littlewood C. Effectiveness of early versus delayed rehabilitation following rotator cuff repair: Systematic review and meta-analyses. PLoS One. 2021 May 28;16(5):e0252137. doi: 10.1371/journal.pone.0252137. eCollection 2021. PMID 34048450
- [Background] Mazuquin BF, Wright AC, Russell S, Monga P, Selfe J, Richards J. Effectiveness of early compared with conservative rehabilitation for patients having rotator cuff repair surgery: an overview of systematic reviews. Br J Sports Med. 2018 Jan;52(2):111-121. doi: 10.1136/bjsports-2016-095963. Epub 2016 Dec 30. PMID 28039127
- [Background] Tirefort J, Schwitzguebel AJ, Collin P, Nowak A, Plomb-Holmes C, Ladermann A. Postoperative Mobilization After Superior Rotator Cuff Repair: Sling Versus No Sling: A Randomized Prospective Study. J Bone Joint Surg Am. 2019 Mar 20;101(6):494-503. doi: 10.2106/JBJS.18.00773. PMID 30893230
- [Background] Ladermann A, Denard PJ, Burkhart SS. Revision arthroscopic rotator cuff repair: systematic review and authors' preferred surgical technique. Arthroscopy. 2012 Aug;28(8):1160-9. doi: 10.1016/j.arthro.2012.01.006. Epub 2012 Apr 6. PMID 22483734
- [Background] Papalia R, Franceschi F, Zampogna B, D'Adamio S, Maffulli N, Denaro V. Augmentation techniques for rotator cuff repair. Br Med Bull. 2013;105:107-38. doi: 10.1093/bmb/lds029. Epub 2012 Oct 18. PMID 23080417
- [Background] Chan K, MacDermid JC, Hoppe DJ, Ayeni OR, Bhandari M, Foote CJ, Athwal GS. Delayed versus early motion after arthroscopic rotator cuff repair: a meta-analysis. J Shoulder Elbow Surg. 2014 Nov;23(11):1631-9. doi: 10.1016/j.jse.2014.05.021. Epub 2014 Aug 13. PMID 25127908
- [Background] Chang KV, Hung CY, Han DS, Chen WS, Wang TG, Chien KL. Early Versus Delayed Passive Range of Motion Exercise for Arthroscopic Rotator Cuff Repair: A Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2015 May;43(5):1265-73. doi: 10.1177/0363546514544698. Epub 2014 Aug 20. PMID 25143489
- [Background] Sheps DM, Silveira A, Beaupre L, Styles-Tripp F, Balyk R, Lalani A, Glasgow R, Bergman J, Bouliane M; Shoulder and Upper Extremity Research Group of Edmonton (SURGE). Early Active Motion Versus Sling Immobilization After Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Arthroscopy. 2019 Mar;35(3):749-760.e2. doi: 10.1016/j.arthro.2018.10.139. PMID 30827428
- [Background] Corban J, Shah S, Ramappa AJ. Current Evidence Based Recommendations on Rehabilitation following Arthroscopic Shoulder Surgery: Rotator Cuff, Instability, Superior Labral Pathology, and Adhesive Capsulitis. Curr Rev Musculoskelet Med. 2024 Jul;17(7):247-257. doi: 10.1007/s12178-024-09899-7. Epub 2024 Apr 26. PMID 38668940
- [Background] Wolf EM, Pennington WT, Agrawal V. Arthroscopic rotator cuff repair: 4- to 10-year results. Arthroscopy. 2004 Jan;20(1):5-12. doi: 10.1016/j.arthro.2003.11.001. PMID 14716273
- [Background] Galatz LM, Griggs S, Cameron BD, Iannotti JP. Prospective longitudinal analysis of postoperative shoulder function : a ten-year follow-up study of full-thickness rotator cuff tears. J Bone Joint Surg Am. 2001 Jul;83(7):1052-6. PMID 11451975
- [Background] Kartus J, Kartus C, Rostgard-Christensen L, Sernert N, Read J, Perko M. Long-term clinical and ultrasound evaluation after arthroscopic acromioplasty in patients with partial rotator cuff tears. Arthroscopy. 2006 Jan;22(1):44-9. doi: 10.1016/j.arthro.2005.07.027. PMID 16399460
- [Background] Weber SC. Arthroscopic debridement and acromioplasty versus mini-open repair in the treatment of significant partial-thickness rotator cuff tears. Arthroscopy. 1999 Mar;15(2):126-31. doi: 10.1053/ar.1999.v15.0150121. PMID 10210067
- [Background] Petersen SA, Murphy TP. The timing of rotator cuff repair for the restoration of function. J Shoulder Elbow Surg. 2011 Jan;20(1):62-8. doi: 10.1016/j.jse.2010.04.045. Epub 2010 Aug 1. PMID 20675154
- [Background] Mantone JK, Burkhead WZ Jr, Noonan J Jr. Nonoperative treatment of rotator cuff tears. Orthop Clin North Am. 2000 Apr;31(2):295-311. doi: 10.1016/s0030-5898(05)70149-8. PMID 10736398
- [Background] Safran O, Schroeder J, Bloom R, Weil Y, Milgrom C. Natural history of nonoperatively treated symptomatic rotator cuff tears in patients 60 years old or younger. Am J Sports Med. 2011 Apr;39(4):710-4. doi: 10.1177/0363546510393944. Epub 2011 Feb 10. PMID 21310940
- [Background] Maman E, Harris C, White L, Tomlinson G, Shashank M, Boynton E. Outcome of nonoperative treatment of symptomatic rotator cuff tears monitored by magnetic resonance imaging. J Bone Joint Surg Am. 2009 Aug;91(8):1898-906. doi: 10.2106/JBJS.G.01335. PMID 19651947
- [Background] Mall NA, Kim HM, Keener JD, Steger-May K, Teefey SA, Middleton WD, Stobbs G, Yamaguchi K. Symptomatic progression of asymptomatic rotator cuff tears: a prospective study of clinical and sonographic variables. J Bone Joint Surg Am. 2010 Nov 17;92(16):2623-33. doi: 10.2106/JBJS.I.00506. PMID 21084574
- [Background] Yamaguchi K, Tetro AM, Blam O, Evanoff BA, Teefey SA, Middleton WD. Natural history of asymptomatic rotator cuff tears: a longitudinal analysis of asymptomatic tears detected sonographically. J Shoulder Elbow Surg. 2001 May-Jun;10(3):199-203. doi: 10.1067/mse.2001.113086. PMID 11408898
- [Background] Tashjian RZ. Epidemiology, natural history, and indications for treatment of rotator cuff tears. Clin Sports Med. 2012 Oct;31(4):589-604. doi: 10.1016/j.csm.2012.07.001. Epub 2012 Aug 30. PMID 23040548
- [Background] Sealey, P. and Lewis, J. (2016) 'Rotator cuff tears: is non-surgical management effective?', Physical Therapy Reviews, 21(3-6), pp. 215-221. doi: 10.1080/10833196.2016.1271504.
- [Background] Flatow EL, Soslowsky LJ, Ticker JB, Pawluk RJ, Hepler M, Ark J, Mow VC, Bigliani LU. Excursion of the rotator cuff under the acromion. Patterns of subacromial contact. Am J Sports Med. 1994 Nov-Dec;22(6):779-88. doi: 10.1177/036354659402200609. PMID 7856802
- [Background] Largacha M, Parsons IM 4th, Campbell B, Titelman RM, Smith KL, Matsen F 3rd. Deficits in shoulder function and general health associated with sixteen common shoulder diagnoses: a study of 2674 patients. J Shoulder Elbow Surg. 2006 Jan-Feb;15(1):30-9. doi: 10.1016/j.jse.2005.04.006. PMID 16414466
- [Background] Carr AJ, Cooper CD, Campbell MK, Rees JL, Moser J, Beard DJ, Fitzpatrick R, Gray A, Dawson J, Murphy J, Bruhn H, Cooper D, Ramsay CR. Clinical effectiveness and cost-effectiveness of open and arthroscopic rotator cuff repair [the UK Rotator Cuff Surgery (UKUFF) randomised trial]. Health Technol Assess. 2015 Oct;19(80):1-218. doi: 10.3310/hta19800. PMID 26463717
- [Background] Cadogan A, Laslett M, Hing WA, McNair PJ, Coates MH. A prospective study of shoulder pain in primary care: prevalence of imaged pathology and response to guided diagnostic blocks. BMC Musculoskelet Disord. 2011 May 28;12:119. doi: 10.1186/1471-2474-12-119. PMID 21619663
- [Background] van der Heijden GJ. Shoulder disorders: a state-of-the-art review. Baillieres Best Pract Res Clin Rheumatol. 1999 Jun;13(2):287-309. doi: 10.1053/berh.1999.0021. PMID 10952865
- [Background] Chester R, Shepstone L, Daniell H, Sweeting D, Lewis J, Jerosch-Herold C. Predicting response to physiotherapy treatment for musculoskeletal shoulder pain: a systematic review. BMC Musculoskelet Disord. 2013 Jul 8;14:203. doi: 10.1186/1471-2474-14-203. PMID 23834747